CLINICAL TRIAL: NCT03038906
Title: Effect of Randomization to Neuromuscular Blockade on Physical Functional Impairment and Recovery in ARDS
Acronym: PRIMROSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Catherine Hough, Associate Professor of Medicine, University of Washington
Other Study IDs: PRIMROSE
Record Dates: First submitted 2017-01-09; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Acute Respiratory Distress Syndrome; Neuromyopathies
MeSH Terms: conditions — Respiratory Distress Syndrome; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Patients enrolling in NHLBI PETAL Network ROSE study of cisatracurium for moderate/severe ARDS at participating centers

SUMMARY:
The proposed work will determine the effect of neuromuscular blockade on physical function and recovery in patients with ARDS. The investigators will conduct a prospective ancillary study at five PETAL clinical centers that will evaluate the neuromuscular structure and function of ROSE (Reevaluation of Systemic Early Neuromuscular Blockade) patients during and after critical illness, including in-person assessments at 6 months after hospital discharge. The investigators hypothesize that patients randomized to NMB will have an increase in ICU-acquired neuromuscular dysfunction during and after critical illness.

DETAILED DESCRIPTION:
The investigators will assess this dysfunction in different ways, appropriate for patients' stage of critical illness and anticipated recovery. During critical illness, the investigators will use nerve conduction studies (NCS) to assess nerve and muscle function, identifying presence of early neuromyopathy (primary outcome, Aim 1). Additional early assessments will include bedside ultrasound to determine muscle mass and echogenicity, indices of atrophy and loss of muscle architecture. Later in acute hospitalization as patients are able to participate in testing, the investigators will use hand grip dynamometry to assess muscle strength (primary outcome, Aim 2). Additional assessments at this time will be hand held dynamometry to determine proximal muscle strength, dual energy x-ray absorptiometry (DEXA) and repeat ultrasound to evaluate muscle mass, and short physical performance battery (SPPB) to assess activity. After hospital discharge-at 6 months after ARDS-the investigators will assess activity in-person using the SPPB (primary outcome, Aim 3). Additional post-hospital assessments include detailed evaluation of healthcare utilization, six minute walk testing (6MWT) to determine endurance, and repetition of previous assessments of muscle structure, function and strength to provide novel, detailed information of recovery process.

Each aim tests a distinct hypothesis of the effect of randomization to NMB on ICU-acquired neuromuscular dysfunction, investigating different time points and aspects of physical function, so aims are not interdependent. For example, it is plausible that the direct toxicity of NMB on muscle will lead to early evidence of neuromyopathy, manifest as reduced muscle depolarization amplitudes with nerve stimulation. But if NMB attenuates lung injury, strength may be improved by hospital discharge, despite early injury to muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled in the PETAL Network's ROSE study
* Patients must have at least one complete leg

Exclusion Criteria:

* Complete spinal cord injury with deficits at level T1 or above
* Severe peripheral neuromuscular disease (specifically motor neuron disease (ALS) or acute Guillain-Barre Syndrome)
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled in the PETAL Network's ROSE (Reevaluation of Systemic Early Neuromuscular Blockade) Study.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Neuromyopathy | Through 6 months after hospital discharge
  The investigators are assessing neuromyopathy with electrophysiologic testing
Muscle Function and Strength | Through 6 months after hospital discharge
  The investigators are assessing muscle strength with handgrip and handheld dynamometry
Physical Recovery and Healthcare Utilization | 6 months post ARDS
  The investigators are assessing physical recovery with the short physical performance battery

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Hough, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No